CLINICAL TRIAL: NCT07209449
Title: Phase II Study of ELacestrant in Combination With Abemaciclib or Elacestrant Alone In p53 Wild Type, Estrogen Receptor-positive Advanced or recurrenT Endometrial Cancer (ELITE)
Brief Title: A Study of Elacestrant Alone or in Combination With Abemaciclib in People With Endometrial Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-164
Record Dates: First submitted 2025-10-01; First posted 2025-10-07 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Cancer
Keywords: Elacestrant; Abemaciclib; p53 Wild Type; Estrogen Receptor-positive; Advanced or Recurrent; 25-164
MeSH Terms: conditions — Endometrial Neoplasms; Recurrence | interventions — abemaciclib; elacestrant

STUDY DESIGN:
Intervention Model Description: This is a phase 2 single institution parallel two-arm randomized trial
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abemaciclib plus Elacestrant (Experimental): Patients receiving both drugs should take elacestrant orally once daily with abemaciclib orally in the morning and abemaciclib orally only in the evening at the same time every day.
  Interventions: Drug: Abemaciclib; Drug: Elacestrant
- Elacestrant alone (Experimental): Patients receiving elacestrant only should take orally once daily in the morning.
  Interventions: Drug: Elacestrant

INTERVENTIONS:
Drug: Abemaciclib — orally only in the evening
  Arms: Abemaciclib plus Elacestrant
Drug: Elacestrant — orally once daily in the morning

SUMMARY:
The researchers are doing this study to find out whether elacestrant is an effective and safe treatment alone or in combination with abemaciclib for people with advanced or recurrent ER+ endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Patients must have received previous platinum-based chemotherapy and treatment with a PD-1 inhibitor, together or separately, prior to enrolling on this trial.
* Patients may have received no more than 1 prior line of chemotherapy for management of endometrial carcinoma. This includes platinum-based chemotherapy alone or combined with a PD-1 inhibitor, small molecule agents, and chemotherapy in combination with radiation therapy. A washout period of 14 days is required for chemotherapy °Adjuvant chemotherapy completed ≥ 12 months prior will not be counted toward prior therapy
* Patients may have received ≤ one prior line of endocrine therapy for management of endometrial carcinoma.
* No prior treatment with a CDK4/6 inhibitor
* Measurable disease per RECIST v 1.1 criteria

  °Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented, or a biopsy is obtained to confirm persistence of tumor ≥ 90 days following completion of radiation therapy.
* Advanced or recurrent endometrial carcinoma that is refractory to curative therapy.
* Patients with the following histologic epithelial cell types are eligible: endometrioid adenocarcinoma, serous adenocarcinoma, undifferentiated carcinoma, de-differentiated, clear cell adenocarcinoma, mixed epithelial carcinoma, adenocarcinoma not otherwise specified (N.O.S.), mucinous adenocarcinoma, squamous cell carcinoma, and transitional cell carcinoma.
* Patient must have ER-positive tumor status either from the most recent sample of advanced/recurrent disease or from an archival tissue.

  °Documentation of ER-positive tumor with ≥ 1% staining by IHC as defined in the 2010 or 2020 American Society for Clinical Oncology recommendations for ER testing (Hammond 2010, Allison 2020)
* p53 wt by IHC or TP53 wt by next generation sequencing platform either from the most recent sample of advanced/recurrent disease or from an archival tissue.
* No known dMMR or POLE mutation
* If MSK IMPACT mutational profiling or mutational profiling performed in a CLIA laboratory is not already performed, must have tissue available for MSK IMPACT molecular profiling to be performed clinically
* Female patients may be either postmenopausal or premenopausal or perimenopausal. Postmenopausal status is defined by:

  * Age ≥ 60 years
  * Age < 60 years and amenorrhea for ≥12 months (in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression) or a follicle-stimulating hormone value >40 mIU/mL and an estradiol value <40 pg/mL or in postmenopausal ranges per local reference ranges
  * Documentation of prior bilateral oophorectomy, at least 1 month before first dose of trial therapy.
  * Premenopausal or perimenopausal patients must be concurrently given a luteinizing hormone-releasing hormone (LHRH) agonist for ovarian suppression starting at least 4 weeks before the start of trial therapy and continue LHRH agonist during the study.
* The effects of elacestrant and abemaciclib on the developing human fetus are unknown. For this reason and because SERDs and CDK4/6 inhibitors as well as other therapeutic agents used in this trial are known to be teratogenic, participants of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) within 28 days of the first dose of study therapy, during study therapy, and for 120 days following the completion of study therapy. Should a participant become pregnant or suspect pregnancy while participating in this study, they should inform their treating physician immediately

  °Highly effective and low user dependency, non-hormonal contraception methods include: i. Intrauterine device (non-hormonal). ii. Total abstinence iii. Bilateral tubal occlusion/ligation. iv. Have a vasectomized partner (sole sexual partner) with confirmed azoospermia
* Any prior radiotherapy directed at the malignant tumor must be discontinued prior to first study treatment. Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between the end of radiotherapy and randomization.
* Have adequate laboratory values as defined below:

  °Hematologic
* Absolute neutrophil count ≥1500/mm3 (≥1.5 × 10^3/μL)
* Platelets ≥100,000/μL
* Hemoglobin ≥9.0 g/dL

  °Renal
* Creatinine clearance (CrCL) Creatinine clearance (CrCl) ≥ 50 mL/min using the Cockcroft-Gault formula

  °Hepatic
* Total bilirubin ≤1.5 ×ULN (patients with known Gilbert's disease who have bilirubin level ≤ 3 x ULN may be enrolled)
* AST and ALT ≤2.5 × ULN (≤5 × ULN for participants with liver metastases)
* Coagulation Prothrombin time (PT) or international normalized ratio (INR) ≤ 1.5 x ULN, and partial prothrombin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN (unless abnormalities are unrelated to coagulopathy or due to prophylactic coagulation)
* Serum Albumin Serum albumin ≥3.0 g/dL (≥30 g/L)

Exclusion Criteria:

* Patient has received an experimental treatment in a clinical trial within the last 30 days or 5 half-lives, whichever is longer, prior to randomization, or is currently enrolled in any other type of medical research not scientifically or medically compatible with this study.
* Patient who is experiencing a visceral crisis, lymphangitic disease spread, leptomeningeal carcinomatosis. Visceral crisis is not the mere presence of visceral metastases but implies severe organ dysfunction as assessed by symptoms and signs, laboratory studies, and rapid progression of disease.
* Patients who have received prior treatment with elacestrant or other investigational oral SERD, everolimus, temsirolimus, ridaforolimus or another mTOR inhibitor, or any CDK4 and CDK6 inhibitor
* Patients with hyperlipidemia that is not adequately controlled.
* Patients with history of interstitial lung disease (ILD)/pneumonitis or evidence of ILD/pneumonitis on baseline imaging.
* Uncontrolled significant active infections. °HIV-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.

control). Patients with a history of treated CNS metastases are eligible, provided that they meet all of the following criteriaFor patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.

* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.

  * Females who are pregnant or nursing. If with childbearing potential, should have a negative urine pregnancy test at the time of screening.
  * Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen.
  * Major surgery within 4 weeks of randomization
  * Inability to take oral medication, or history of malabsorption syndrome or any other uncontrolled gastrointestinal condition.
  * Known intolerance to either study drug or any of the excipients.
  * Any severe medical or psychiatric condition that in the opinion of the investigator(s) would preclude the patient's participation in a clinical study.
  * Uncontrolled hypomagnesemia or hypokalemia, defined as values below the lower limit of normal despite optimal electrolyte supplementation or management
  * Known untreated or active central nervous system (CNS) metastases (progression or requiring anticonvulsants or corticosteroids for symptomatic control). Patients with a history of treated CNS metastases are eligible, provided that they meet all of the following criteria:
* Presence of measurable disease outside the CNS
* No radiographic evidence of worsening upon the completion of CNS-directed therapy and no evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study
* No history of intracranial hemorrhage or spinal cord hemorrhage
* No ongoing requirement for dexamethasone as therapy for CNS disease (anticonvulsants at a stable dose are allowed)
* Screening CNS radiographic study is within 6 months after most recent intervention for CNS metastases and greater than 4 months after discontinuation of corticosteroids

  * Inability to comply with study and follow-up procedures
  * Patient is currently receiving or received any of the following medications prior to first dose of trial therapy:
* Known strong or moderate inducers or inhibitors of cytochrome P450 (CYP) 3A4 (including foods and herbal preparations) within 14 days or 5 half-lives, whichever is shorter, prior to initiating study therapy.
* Herbal preparations/medications. These include, but are not limited to, St.John's wort, kava, ephedra (ma huang), ginkgo biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng within 21 days prior to initiating trial therapy

  * Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Endometrial Cancer
Enrollment: 75 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2028-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 1 year
  according to RECIST 1.1 criteria. Defined as the percentage of patients with complete response (CR) + partial response (PR)] after initiating therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Green, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/